CLINICAL TRIAL: NCT04865796
Title: Epidemiology, Clinical Evaluation of Black Stains and Patients' Dietary Habits: a Clinical Trial.
Brief Title: Black Stains' Epidemiology, Clinical Evaluation and Dietary Habits: a Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Research Resident, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-BLACKSTAINS
Record Dates: First submitted 2021-04-26; First posted 2021-04-29 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Black Stains
Keywords: Oral microbiota; Periodontal bacteria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Experimental): Patients will use products based on lactoferrin.
  Interventions: Other: Lactoferrin products
- Probiotics (Experimental): Patients will use products based on probiotics for home oral care.
  Interventions: Other: Probiotics products
- Standard therapy (Active Comparator): Patients will use standard toothpastes for home oral care.
  Interventions: Other: Standard home oral care

INTERVENTIONS:
Other: Lactoferrin products — Patiens will use a toothpaste and 2 tablets per day (between foods) for home oral care.
  Arms: Group 1
Other: Probiotics products — Patiens will use a toothpaste and a chewing-gum (for 10 minutes a day) for home oral care.
  Arms: Probiotics
Other: Standard home oral care — Patiens will use a normal toothpaste for home oral care.
  Arms: Standard therapy

SUMMARY:
The aim of this study is to investigate epidemiology and treatment possibilities of black stains, with the assessment of a possible correlation with patients' dietary habits.

Patients will be randomly divided into three groups. For each group, clinical evaluation will be performed at the study begin, after 2 and after 6 months.

At the study begin, evaluation of black stains with Gasparetto's classification will be assessed; then professional oral hygiene with ultrasonic scaler will be performed, plus glycine and polish; then, products for home oral care will be given to patients, depending on the groups. The clinical situation will be re-evaluated after 2 and after 6 months. Home oral care will be performed with different products, containing lactoferrin (group 1) and probiotics (group 2). The control group (Group 3) will use normal products.

DETAILED DESCRIPTION:
The aim of this study is to investigate epidemiology and treatment possibilities of black stains, with the assessment of a possible correlation with patients' dietary habits.

Patients will be randomly divided into three groups. For each group, clinical evaluation will be performed at the study begin, after 2 and after 6 months.

At the study begin, evaluation of black stains with Gasparetto's classification will be assessed; then professional oral hygiene with ultrasonic scaler will be performed, plus glycine and polish; then, products for home oral care will be given to patients, depending on the groups. The clinical situation will be re-evaluated after 2 and after 6 months.

Home oral care will be performed as follows:

* Group 1: patients will use 2 Forhans GengiFor tables (between foods) and Forhans Scudo Naturale toothpaste containing lactoferrin.
* Group 2: patients will use Biorepair Peribioma chewing-gum for 10 minutes/day and Biorepair Peribioma toothpaste containing probiotics.
* Group 3: patients will choose the best product for their home oral care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with black stains
* Patients with high compliance

Exclusion Criteria:

* Patients suffering from psychological, neurological or psychiatric disorders
* Pregnant or breastfeeding women
* Patients undergoing anti-cancer therapy
* Patients with low compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-05-15 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-16 (Actual)

PRIMARY OUTCOMES:
Change in the extension of black stains (Gasparetto et al., 2003) | Study begin, 2 and 6 months.
  Scoring criteria:
  * 1: presence of pigmented dots or thin lines with incomplete coalescence parallel to gingival margin;
  * 2: continuous pigmented lines, which can be easily observed and limited to half of the cervical third of the tooth surface;
  * 3: presence of pigmented stains extending beyond half of the cervical third of the tooth surface

SECONDARY OUTCOMES:
Change in DMFT (Decayed Missing Filled Teeth) score | Study begin, 2 and 6 months.
  It's the measure of caries experience worldwide. This index gives the sum of an individual's decayed, missing, and filled permanent teeth. It ranges from 0 to 32 (including the wisdom teeth). The higher the score, the worst the oral health condition of the patient.
Change in DMFS (Decayed Missing Filled Surfaces) score | Study begin, 2 and 6 months.
  It's the measure of caries experience worldwide. This index gives the sum of an individual's decayed, missing, and filled permanent surfaces. It ranges from 0 to 148 (including the wisdom teeth). The higher the score, the worst the oral health condition of the patient.
Dietary habits | Study begin, 2 and 6 months.
  Patients will ask to assess if there is a consumption of the following foods and drinks ≤ 3 times /months, ≤ 6/week, ≥ 1/day:
  Beet Swiss chard Broccoli Candies Meat Cabbage Desserts Fresh fruit Dairy product Legumes Spinach Eggs Vegetable Coffee Coca Cola Natural juices Red juices The Red wine

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD., Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator